CLINICAL TRIAL: NCT04811196
Title: A Phase 1 Study of Metronomic Selinexor in Select Soft Tissue Sarcomas and Split Dosing of Selinexor in All Soft Tissue Sarcomas
Brief Title: A Study of Different Dosing Schedules of Selinexor in Sarcoma Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: METSSAR
Record Dates: First submitted 2021-01-25; First posted 2021-03-23 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Soft Tissue Sarcoma; Malignant Peripheral Nerve Sheath Tumor (MPNST); Leiomyosarcoma; Endometrial Stromal Sarcoma
Keywords: Selinexor, Sarcoma
MeSH Terms: conditions — Sarcoma; Neurofibrosarcoma; Leiomyosarcoma; Sarcoma, Endometrial Stromal | interventions — selinexor

STUDY DESIGN:
Intervention Model Description: This is a phase 1/1b single centre study with two arms. Arm A is a dose escalation study assessing the safety, tolerability and preliminary antitumor activity of low dose metronomic Selinexor in adult patients with locally advanced/unresectable or metastatic MPNST, endometrial stromal cell sarcomas or angiogenic tumors. This is a dose escalation study and will consist of ascending doses of Selinexor administered metronomically as a single agent.
  Up to 36 patients will be enrolled in Arm A.
  Arm B of this study will enroll all soft tissue sarcoma histologies to receive flat dosing Selinexor 40mg in the morning, 20mg in the afternoon and 20mg at night orally on days 1, 8, 15, 22 of a 28-day cycle. Twenty patients will be enrolled to this arm. This pattern will continue until disease progression or unacceptable toxicity. Quality of life assessments will occur at pre-dosing, cycle 2 day 1, cycle 6 day 1 and cycle 12 day 1 for those who remain on study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Metronomic dosing (Experimental): This Arm is an open-label, non-randomized, phase 1 study of metronomic dosing of selinexor in patients with locally advanced or metastatic MPNST, ESS, LMS. Up to seven dose levels of Selinexor will be investigated.
  Patients will undergo 3+3 based dose escalation to determine the maximum tolerated dose (MTD) and recommended phase 2 dose (RP2D) of Selinexor.
  Escalating doses of selinexor will be given starting with 2.5 mg (taken orally 4 days in a row followed by 3 days break from treatment, repeating this weekly as part of a 28-day cycle). The first dose for the first 2 patients at each dose level will be staggered by 7 days. Minimum number of patients treated in this trial arm is 18 patients, and maximum 36 patients.
  Schedule:
  Selinexor flat dosing with dose levels (DLs) of 2.5mg (DL1), 5mg (DL2), 7.5mg (DL3), 10mg (DL4), 12.5mg (DL5), 15mg (DL6), 17.5mg (DL7). A DL-1 (1.25 mg) is also incorporated.
  Interventions: Drug: Selinexor
- Split dosing (Experimental): The second arm of the study is an open-label, non randomized, phase 1b study of selinexor in patients with any histological subtype of STS administered orally one day per week, 40mg in the morning, 20mg in the afternoon and 20mg at night as part of a 28 day cycle. Twenty patients will be accrued to this arm.
  Interventions: Drug: Selinexor

INTERVENTIONS:
Drug: Selinexor — Selinexor
  Other Names: KPT-330, XPOVIO

SUMMARY:
This is a phase 1, open-label, single centre study of investigational drug selinexor in participants with soft tissue sarcomas that cannot be treated with standard therapies. Selinexor has been given to 3111 participants with cancer to date including 142 sarcoma patients. Early findings have shown that selinexor is effective in multiple cancer types. The current study is being done to test low doses and different dosing schedules of selinexor to find out if it reduces the side effects without compromising the benefits.

This study has 2 groups or Arms: Arm A and Arm B.

Arm A (Dose escalation Arm): Participants will receive selinexor by mouth 4 days a week to find out the safety, tolerability and anti-tumor effect of low doses of Selinexor in participants with advanced or metastatic malignant peripheral nerve sheath tumors (MPNST), endometrial stromal sarcomas (ESS) and leiomyosarcoma (LMS). Participants will continue on study until disease progression or unacceptable side effects. Up to 36 participants will be enrolled in this Arm.

Arm B: Participants with any soft tissue sarcoma subtypes will be enrolled in this Arm. They will receive flat doses of Selinexor by mouth once weekly, 3 times a day. Safety and tolerability will be assessed in this Arm. Up to 20 participants will be enrolled and they will continue to receive selinexor until disease progression or unacceptable side effects.

Cancer is the uncontrolled growth of human cells. One of the ways cancers cells continue to grow is by getting rid of proteins called "tumor suppressor proteins" that would normally cause cancer cells to die. The study drug works by trapping "tumor suppressor proteins" within the cell, causing the cancer cells to die or stop growing.

The study comprises 3 periods: Screening (up to 28 days), Study Drug (until disease progression), and Survival Follow-Up (once every 3 months). Procedures for research purposes only will include blood collection and study questionnaire.

DETAILED DESCRIPTION:
Background:

Soft tissue sarcomas (STS):

STS are a group of heterogeneous mesenchymal derived tumors with many histological types that account for approximately 1% of adult tumors and 15% of pediatric tumors. STS can be divided into those with simple genetic alterations (e.g. translocations or activating mutations) or karyotypic complex lesions. However, most subclasses are treated in the same manner. Surgery is the primary treatment for localized STS, with or without radiation therapy (RT), but approximately 10% of patients will present with metastatic disease.

For patients who present with metastatic disease, or those with locally advanced/unresectable or have failed primary therapy, cytotoxic chemotherapy is usually the treatment of choice which may provide meaningful palliation or prolong survival. Traditionally, doxorubicin containing regimens, in combination with ifosfamide or as a single agent are standard first line therapies. Combination based doxorubicin containing regimens have shown higher response rates and progression free survival at the expense of more toxicity when compared to doxorubicin alone. However, no combination regimen has been associated with increased overall survival compared to doxorubicin alone.

In the metastatic setting, STS carry a poor prognosis related to a lack of chemo-sensitivity and a lack of systemic therapeutic options. Exportin 1 (XPO1 or chromosome region maintenance 1 [CRM1]) is the sole nuclear exporter of some tumor suppressor proteins (TSP). XPO1 is over-expressed 2-4 fold in a variety of solid and hematological tumors with higher levels correlating with poorer outcomes.

Selinexor:

Selinexor is a novel, oral, small-molecule XPO1 inhibitor which forces reactivation of TSPs and thus leads to apoptosis of tumor cells. Preclinical data of Selinexor has shown promising in-vitro tumor regression in sarcoma. In two phase I studies, single agent clinical activity in the form of prolonged stable disease was seen in STS. Twice weekly dosing aided tolerability with a MTD declared at 65mg/m2 for solid tumors and 60mg flat dosing was the RP2D based on better tolerability given problems related to gastrointestinal toxicity however these doses were still difficult for patients to take due to the toxicity profile. A Phase 1b study has been performed combining Selinexor once weekly oral dosing with doxorubicin given at the standard 3 weekly dose in advanced soft tissue sarcoma.

Previous studies have provided a signal of increased likelihood of benefit to particular subtypes including metastatic malignant peripheral nerve sheath tumors (MPNST) and endometrial stromal sarcomas (ESS). In the early phase studies, objective responses or prolonged stable disease were demonstrated (n=3 for both MPNST and ESS). In this study, the investigator also plans to include leiomyosarcoma (LMS) - such strategy will allow not only seamless recruitment, but also generate treatment efficacy data for other rare types of sarcomas.

Additionally, preclinical data has shown efficacy in using metronomic dosing of Selinexor. The investigator hypothesizes that low dose Selinexor will improve tolerability of the drug without impacting the clinical benefit that has been seen in other studies for patients with particular histological subtypes of STS.

Rationale:

Biological Rationale:

More than 2500 patients with advanced cancers have received Selinexor orally in Phase 1 and Phase 2-3 studies as of 31 May 2019. Based on the preclinical and clinical findings to date, Selinexor dosing is limited to ≤70 mg/m2 (≤120 mg) maximum dose in adults. The plan going forward is that Selinexor will be administered primarily as fixed milligram doses, as analyses of Phase 1 pharmacokinetic (PK) data indicated that exposure is not strongly correlated with Body Surface Area (BSA).

An interim analysis of preliminary results was performed to determine the RP2D for future studies. The results of this analysis suggest that, overall, Selinexor doses > 65 mg do not appear to provide additional efficacy responses beyond those seen with the 60 mg dose (described herein as 45-65 mg dose level, median 60 mg) with the exception of activity in refractory multiple myeloma (MM), where the RP2D is Selinexor 80 mg in combination with 20mg dexamethasone. Importantly, response results with Selinexor 45-65 mg twice weekly were comparable for both hematologic malignancies (excluding MM) and solid tumors.

The currently available selinexor formulation (20 mg tablet) and dosage is quite toxic particularly in terms of gastrointestinal disturbance, particularly nausea and vomiting. As a result of these difficulties it might be beneficial to investigate alternate formulations of selinexor or a different dosing schedule of the currently available selinexor formulation. A PK study in male Beagle dogs has been completed by Karyopharm investigating a new extended release (ER) formulation of Selinexor 20 mg tablets showing favorable results.

Dose Schedule Rationale:

In the present study, Selinexor will be given using two different schedules according to Schema for Arm A (metronomic) and Schema for Arm B (split dosing).

In Arm A Selinexor will be administered at a fixed oral dose as per dose level (starting at 2.5mg PO 4 days on, 3 days off repeated weekly) of each 4-week (28-day) cycle a total of 16 doses per cycle. The maximum dose for Selinexor in this study will be 17.5mg PO flat dosing 4 days on, 3 days off, weekly. This arm of the study will be aimed at identifying the RP2D and toxicity profile of this new selinexor dosing schedule.

In Arm B patients will be treated with Selinexor 40mg in the morning, 20mg in the afternoon and 20mg at night on days 1, 8, 15 and 22 of a 28-day cycle. The hope is that this alternate dosing schedule will improve the tolerability of this formulation of selinexor without impacting its clinical benefit.

Intervention and mode of delivery:

In Arm A patients will receive Selinexor orally as described above. The initial 3 patients will be enrolled to the first Selinexor dose level of 2.5mg (DL1). Three patients will be assessed per cohort for at least 1 cycle and dose escalation or de-escalation rules will follow 3+3 dosing. The first dose of study treatment for the first two patients will be staggered by 7 days. Intra-patient dose escalation is not permitted at any time during the treatment plan.

In Arm B also patients will receive selinexor orally as described above.

Duration of Intervention and Evaluation:

Treatment in both arms with Selinexor will be repeated on a 28-day cycle until radiographic or symptomatic progression on imaging or the development of unacceptable toxicity. Patients will be restaged every 2 cycles until unacceptable toxicity or disease progression. Subsequent follow-up for disease progression will continue by telephone or review of patient medical records for up to 2 years after the completion of trial treatment.

Number of Patients:

A total of up to 36 patients will be accrued in Arm A. Up to 20 patients will be enrolled in Arm B with an anticipated accrual period of 12 to 18 months.

Definition of dose limiting toxicity (DLT):

DLT is defined as any of the following occurring in the first 28 days of each dose level that is considered at least possibly related to drug administration:

≥ 4 missed doses (out of 16) due to a toxicity that is at least possibly study drug related.

Discontinuation of a patient due a toxicity that is at least possibly study drug related before completing cycle 1

Non-Hematologic:

Grade ≥ 3 nausea/vomiting, dehydration or diarrhea while taking optimal supportive medications Grade 3 fatigue lasting for ≥ 7 days while taking optimal supportive care and with correction of dehydration, anorexia, anemia, endocrine, or electrolyte abnormalities.

Grade 3 AST or ALT elevation lasting longer than 7 days OR Grade 3 AST or ALT elevation in the setting of bilirubin elevation > 2x ULN (> 2X baseline for patients with Gilbert's syndrome) OR any grade 4 AST or ALT elevation.

Any other clinically significant Grade ≥ 3 non-hematological toxicity except alopecia or electrolyte abnormalities correctable with supportive therapy Any cardiac disorder ≥ CTCAE Grade 3

Hematologic:

Grade 4 neutropenia [absolute neutrophil count (ANC) < 0.5x109/L] on Cycle 2 Day 1 that does not resolve to G1 within 7 days Grade 4 neutropenia [absolute neutrophil count (ANC) < 0.5x109/L] within the first 28 days lasting ≥ 7 days Grade 3 Febrile neutropenia Grade ≥ 3 thrombocytopenia associated with clinically significant bleeding Grade 4 thrombocytopenia within the first 28 days (platelets < 25x109/L) lasting > 7days

Other:

Any hematologic or non-hematologic toxicity that results in the inability to administer day 1 of the next planned cycle within 14 days of the planned end of the previous cycle.

Treatment related death During the dose escalation portion of the study, patients who missed >1 dose of Selinexor during Cycle 1 for reasons unrelated to study drug are not evaluable for DLT and will be replaced.

Treatment Discontinuation Criteria:

Disease progression Noncompliance with protocol Need for treatment with medications not allowed by the study protocol Consent withdrawal Intercurrent illness Incidence or severity of AEs Investigator discretion

Duration:

The treatment period for an individual patient is expected to be approximately between 2 and 12 months, however there is no maximum treatment duration.

Study procedures:

For Arm A the starting dose of Selinexor will be 2.5mg given 4 days on 3 days off on a weekly basis as part of a 28-day cycle. For Arm B patients will receive oral Selinexor 40 mg in the morning, 20 mg in the afternoon, 20 mg in the evening. Patients will be assessed for response after ever 2 cycles. Treatment will be given until disease progression or unacceptable toxicity.

Safety data:

Overall safety profile as per NCI CTCAE version 5.

Concomitant Medications:

Patients will receive best supportive care, including anti-emetics, appetite stimulants and growth factors, blood product transfusions, antimicrobials and (as appropriate) granulocyte colony-stimulating factors (G-CSF) for neutropenia and/or neutropenic infection, erythropoietin for anemia, and/or platelet-stimulating factors for thrombocytopenia. Patients will not be dosed with G-CSF in the first cycle for primary prophylaxis of febrile neutropenia.

If clinically indicated and as required by protocol, patients may receive red blood cell or platelet transfusions, acetaminophen, serotonin (5-HT3) receptor subtype antagonists (e.g., ondansetron) megestrol acetate, and olanzapine in addition to ondansetron. Patients intolerant to 5-HT3 antagonists may receive D2-antagonists instead. Additional anti-nausea and anti-anorexia agents may be given as needed. Patients may continue to receive baseline medication(s), and may receive concomitant medications that are medically necessary as standard care to treat co-morbid diseases, AEs, and intercurrent illnesses.

Concurrent therapy with any other approved or investigative anticancer therapy is not allowed.

Pharmacokinetic and Pharmacodynamic assessments:

PK will be determined at various times following administration of Selinexor in Arm A.

Pharmacokinetics:

In the metronomic arm for the first 3 patients in each dose level, blood samples just before Selinexor administration (C1D1), and at 1hr, 2hr, 4hr, 24hr and a trough level pre C2 will be collected.

Response:

Objective disease response assessment will be made according to standard, international RECIST 1.1 criteria for solid tumors.

Safety Variables and Analysis:

The safety and tolerability of Selinexor will be evaluated by means of drug related DLT, AE reports, physical examinations, and clinically significant laboratory safety evaluations. NCI CTCAE version 5.0 will be used for grading of AEs.

Investigators will provide their assessment of causality as: unrelated, possibly related, or probably or definitely related for all AEs.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent in accordance with federal, local, and institutional guidelines
2. Age > 18 years.
3. Patients must have histologically confirmed locally advanced/unresectable or metastatic STS

   1. For Arm A the acceptable histologies are MPNST, ESS and LMS
   2. For Arm B arm all STS histologies are eligible
4. Patients must fall into one of the three following categories:

   1. Show evidence of progressive disease on study entry; or
   2. Be treatment naïve, but have progressed since diagnosis; or
   3. Newly diagnosed patients with de novo metastatic measurable disease.
5. Patient must have measureable disease as defined by RECIST 1.1.
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
7. Adequate hematopoietic function within 7 days prior to C1D1:

   1. absolute neutrophil count (ANC) ≥1.0x109/L
   2. hemoglobin ≥ 90 g/L
   3. platelet count ≥100 x 109/L
   4. Patients receiving hematopoietic growth factor support, including erythropoietin, darbepoetin, granulocyte-colony stimulating factor (G-CSF), granulocyte macrophage-colony stimulating factor (GM-CSF), and platelet stimulators (eg, eltrombopag, romiplostim, or interleukin-11) must have a 2-week interval between growth factor support and the Screening assessments, but they may receive growth factor support during the study.
   5. Patients must have:

   i. At least a 2-week interval from the last red blood cell (RBC) transfusion prior to the Screening hemoglobin assessment, and

   ii. At least a 1-week interval from the last platelet transfusion prior to the Screening platelet assessment.

   iii. However, patients may receive RBC and/or platelet transfusions as clinically indicated per institutional guidelines during the study.
8. Adequate hepatic function within 28 days prior to C1D1:

   1. Bilirubin <1.5 times the upper limit of normal (ULN) (except patients with Gilbert's syndrome who must have a total bilirubin of < 3 times ULN)
   2. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) <2 X ULN. In the case of known (radiological and/or biopsy documented) liver metastasis, ALT/AST <5.0 X ULN is acceptable;
9. Adequate renal function within 28 days prior to C1D1: estimated creatinine clearance of ≥20 mL/min calculated using the formula of Cockcroft and Gault: (140-Age)(Weight in kg)(Constant)/(serum creatinine µmol/L); where constant is 1.23 for men and by 1.04 for women.
10. Female patients of childbearing potential must agree to use two methods of contraception (including one highly effective and one effective method of contraception) and have a negative serum pregnancy test at Screening. Male patients must use an effective barrier method of contraception if sexually active with a female of childbearing potential. For both male and female patients, effective methods of contraception must be used throughout the study and for 3 months following the last dose of study treatment.
11. Ability to swallow pills

Exclusion Criteria:

1. Has received selinexor or another XPO1 inhibitor previously
2. Patients who are pregnant or lactating
3. Radiation (except planned or on-going palliative radiation outside of the region of measurable disease), chemotherapy, immunotherapy, any other systemic anticancer therapy, or participation in an investigational anti-cancer study ≤3 weeks prior to initiation of therapy. Mitomycin C and radio-immunotherapy within 6 weeks prior to cycle 1 day 1.
4. Major surgery within 4 weeks before initiation of therapy
5. Active, ongoing or uncontrolled active infection within one week prior to first dose
6. Patients with any gastrointestinal dysfunctions that could interfere with the absorption of Selinexor or patients with significantly diseased or obstructed gastrointestinal tract or uncontrolled vomiting or diarrhea;
7. Inability or unwillingness to take supportive medications such as anti-nausea and anti anorexia agents as recommended by the National Comprehensive Cancer Network (NCCN) Clinical Practice Guidelines for Antiemesis and Palliative Care.
8. In the opinion of the Investigator, patients who are significantly below their ideal body weight (Body Surface Area ≤ 1.2m2)
9. Concurrent therapy with approved or investigational anticancer therapeutic agents
10. Any condition that, in the opinion of the Investigator, would interfere with evaluation of the study regimen or interpretation of patient safety or study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2021-03-29 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2025-05-15 (Actual)

PRIMARY OUTCOMES:
Incidence of toxicity and safety of Selinexor given on either a metronomic (Arm A) or split dosing (Arm B) schedule: Adverse Events | Up to 14 days after completion of study treatment
  Graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. Analyses will be performed using descriptive statistics.
Recommended phase 2 dose of Selinexor given metronomically | Up to 28 days
  Toxicity will be assessed using the NCI CTCAE, version 5.0. Adverse events will be tabulated and summarized by major organ category, grade, anticipation, and drug attribution.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) of metronomic Selinexor | From date of first dose of selinexor until the date of first documented progression, assessed up to 12 months.
  The Kaplan-Meier product limit method will be used to estimate PFS of the median PFS and PFS rates at clinically relevant time point will be provided with the 95% CI.
Objective Response Rate (ORR) of metronomic Selinexor | From date of first dose of selinexor until the date of first documented progression, assessed up to 12 months.
  Defined as the proportion of patients who achieved a complete response (disappearance of all target tumors) or a partial response (PR) (≥30% decrease in the sum of longest diameters of target tumors) based on RECIST Version 1.1. The ORR, along with exact two-sided 95% confidence intervals based on binomial distribution will be reported.
Clinical Benefit Rate (CBR) of metronomic Selinexor | From date of first dose of selinexor until the date of first documented progression, assessed up to 12 months.
  Defined as the proportion of patients who achieved a complete response (disappearance of all target tumors) or a partial response (≥30% decrease in the sum of the longest diameters of target tumors) or stable disease (Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD) for greater than 16 weeks based on RECIST Version 1.1. The CBR, along with exact two-sided 95% confidence intervals based on binomial distribution will be reported.
Peak Plasma Concentration (Cmax) of metronomic Selinexor | Prior to dose on day 1, and at 1, 2, 4, and 24 hours post dose of Cycle 1, and prior to dose on Day 1 of Cycle 2 (each cycle is 28 days).
  Descriptive statistics will be used to summarize Selinexor concentration at each sampling time point and Cmax. Only the first 3 patients per dose level will be included for Cmax analysis.
Area under the plasma concentration versus time curve (AUC) of metronomic Selinexor | Prior to dose on day 1, and at 1, 2, 4, and 24 hours post dose of Cycle 1, and prior to dose on Day 1 of Cycle 2 (each cycle is 28 days).
  Descriptive statistics will be used to summarize AUC of Selinexor. Only the first 3 patients per dose level will be included for AUC analysis.
Characterization of the toxicity of metronomic Selinexor | Up to 14 days after completion of study treatment
  Analyses will be performed for all patients having received at least one dose of study drug. The study will use the NCI CTCAE v5.0. Serious adverse events, AEs, AEs leading to withdrawal/dose interruptions/dose modification will be summarized using descriptive statistics.
Quality of life assessment using Quality of Life Questionnaire | Screening and then pre-dose Cycles 1, 6, and 12 (each cycle is 28 days).
  To better define the toxicity of Selinexor, patient reported outcomes using 'European Organization for Research and Treatment of Cancer' (EORTC) 'Quality of Life Questionnaire' (QLQ-C30) will be investigated. The score ranges from 1 to 4, with 1 being the worst outcome and 4 being the best. Mean score of individual item numbers of interest will be analyzed with descriptive and mixed effect model methods.

CONTACTS AND LOCATIONS:
Overall Officials: Albiruni Razak, M.D., Principal Investigator — Princess Margaret Cancer Centre
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No